CLINICAL TRIAL: NCT03350373
Title: Clinical Pharmacology Study of Final Formulation of FYU-981 Administered to Healthy Male Adults
Brief Title: Clinical Pharmacology of FYU-981 (Final Formulation)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Collaborators: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-016
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — dotinurad

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted dosing followed by fed dosing (Experimental): Dosing of FYU-981 in the fasted state followed by fed dosing
  Interventions: Drug: FYU-981
- Fed dosing followed by fasted dosing (Experimental): Dosing of FYU-981 in the fed state followed by fasted dosing
  Interventions: Drug: FYU-981

INTERVENTIONS:
Drug: FYU-981 — Single administration of FYU-981 under Fasted and fed conditions in the morning.
  Other Names: Final formulation of FYU-981

SUMMARY:
This is a randomized, open-label, 2-period crossover study. The purpose of this study is to assess the pharmacokinetics and safety after single oral administration of final formulation of FYU-981 to healthy male adults in fasted and fed conditions. Participants are randomized to fasted (n=6) or fed conditions (n=6) in each step. The effect of food to pharmacokinetics of FYU-981 is also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy adult subjects
* Body mass index: >=18.5 and <25.0

Exclusion Criteria:

* Subjects with any disease or any history of diseases that might be unsuitable for participation in the clinical study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 48 hours
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 48 hours
Pharmacokinetics | 48 hours
  T1/2: Elimination half-life of plasma concentration
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 48 hours
Pharmacokinetics (CLtot/F: Total clearance/Fraction of dose absorbed) | 48 hours
Pharmacokinetics (kel: Elimination rate constant) | 48 hours
Pharmacokinetics (Vd/F: Distribution volume/Fraction of dose absorbed) | 48 hours
Pharmacokinetics (MRT: Mean residence time) | 48 hours
Safety (Incidence of treatment-emergent adverse events) | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Katsuaki Nagasawa, Study Director — Clinical Research Department
Locations (1):
- P-One Clinic, Hachiōji, Tokyo, Japan